CLINICAL TRIAL: NCT05676047
Title: Symptom-Targeted Rehabilitation for Cognitive Complaints in Long COVID (STAR-C3)
Brief Title: Cognitive Rehabilitation for Long COVID
Acronym: STAR-C3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15621
Record Dates: First submitted 2023-01-04; First posted 2023-01-09 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Long COVID
Keywords: Cognitive Rehabilitation; Cognitive Functioning
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Cognitive Training; Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the Therapy (n=50) or Education Group (n=50). At the conclusion of therapy (for the Therapy Group) or after three weeks (for the Education Group), participants will be re-administered the outcome measures. The outcome measures using the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) will then be compared during data analysis between the two groups.
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blinded to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapy Group (Experimental): The Therapy Group will receive 6-10 individual sessions of 30-60 minutes each, delivered by a trained Occupational Therapist or Speech-Language Pathologist. The therapy will be delivered over a 4-week timeframe, with the total number of sessions per participant depending on the number of sessions needed to achieve their treatment targets. Each participant in the Therapy Group will identify three cognitive targets for treatment. Progress in reaching those targets will be documented using Goal Attainment Scaling (GAS)
  Interventions: Behavioral: Cognitive Rehabilitation
- Educational Group (Active Comparator): The Education group will receive information about self-management of cognitive symptoms at the time of randomization, a common alternative for adults with Long COVID cognitive symptoms who do not receive Individual Therapy.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — A strategy-focused intervention aimed at improving everyday cognitive function, structured to maximize treatment dose over a short time period. The shorter time period of the treatment therapy is relative to the one and only current randomized controlled trial of cognitive rehabilitation for military mTBI, the Study of Cognitive Rehabilitation Effectiveness (SCORE).
  Arms: Therapy Group
Other: Education — The Education group will receive information about self-management of cognitive symptoms at the time of randomization, a common alternative for adults with Long COVID cognitive symptoms who do not receive Individual Therapy.
  Arms: Educational Group

SUMMARY:
The investigators are comparing two different methods for helping adults with Long Coronavirus (COVID) also known as Post-Coronavirus Syndrome or Post-Coronavirus Condition manage everyday cognitive challenges. Cognitive rehabilitation is a type of therapy that helps people who have challenges with everyday thinking because of a brain injury. One of the investigators on this project along with colleagues in the United States (US) have developed a streamlined version of cognitive rehabilitation therapy for mild traumatic brain injury (mTBI) that can be completed in person or virtually and takes place over a 3-week period. The therapy was originally designed for adults with mTBI. The investigators want to know if it can also be used to treat people with cognitive complaints from Long COVID. The investigators will provide education materials only to one group and individual cognitive rehabilitation delivered by a trained Speech Language Pathologist (SLP) or Occupational Therapist (OT) to the other group. The investigators want to find out whether the individual therapy is as feasible and accessible than the usual educational material. What the investigators learn in this study may help treat day-to-day thinking challenges in Long COVID.

DETAILED DESCRIPTION:
Cognitive complaints are one of the most common, pervasive, and debilitating outcomes for adults with Long COVID. In a study of 3762 adults from 56 countries who were 7 months post-diagnosis of severe acute respiratory syndrome coronavirus-2 (SARS Coronavirus 2, referred to here as COVID) 85% reported cognitive problems, including brain fog, word-finding problems, difficulty communicating their thoughts, and a reduced ability to solve serious problems. In the Great British Intelligence Test, an online study of 81,337 individuals the subgroup of 12,689 who reported having had COVID had significantly lower cognitive test scores than those who had not, providing objective support for the symptoms that adults with Long COVID are reporting. These persistent cognitive symptoms, which the investigators refer to as Post-COVID Cognitive Symptoms (PCCS), do not appear to spontaneously resolve, with many patients in Canada and worldwide reporting cognitive impairments more than 1 year after infection. PCCS can have severe effects on usual functioning, particularly given that most survivors are working age. Two large studies estimated that at 7-9 months post-infection, between 40-75% of adults either could not work at all or were working fewer hours than they did pre-COVID. Although emerging data indicate that PCCS may be less common after infection with the Omicron variant, there continues to be concern about future "super-variants" that may have more virulent effects. Even if infection rates stabilize, i.e., COVID becomes endemic, the disease does not become harmless.

Usual care for those with PCCS is, at best, providing information about how to manage symptoms (e.g., this handout from the Public Health Authority of British Columbia). The literature on treatment of cognitive problems in other patient groups, however, shows that providing general information alone does not "fix" cognitive impairments. To improve cognitive function in everyday life, intervention must be individualized and provide opportunities for high-dose practice of target behaviours. The investigators do not, however, have interventions like this with demonstrated effectiveness for PCCS. The literature related to cognitive rehabilitation after COVID includes three types of papers: 1) studies of COVID effects on people who had cognitive diagnoses pre-COVID (e.g., how lack of services has affected patients with Alzheimer's Disease) 2) a small number of case reports of rehabilitation for COVID patients, in which cognitive rehabilitation is mentioned in general terms (e.g., patient received "skill training for basic activities of living" and "evaluation of adaptive devices", and 3) urgent calls for cognitive rehabilitation of adults with PCCS (e.g., 13-15). To the investigators knowledge, there are no published controlled studies of cognitive rehabilitation methods for adults with PCCS. One of the investigators recently completed a pilot pre-post study with 34 adults with Long COVID to examine if physical therapy for physical symptoms and occupational therapy for cognitive symptoms was safe and feasible (protocol completed, under analysis). The cognitive intervention was 6 hours of combined individual and group cognitive rehabilitation over 12 weeks, including education about managing cognitive challenges. The pilot data showed a reduction in intensity and frequency of cognitive symptoms, but no effect on everyday functioning. The study investigators concluded that to improve everyday function, therapy must be targeted at individual complaints, and it is this type of intervention that the investigators propose for a randomized control trial (RCT).

A recent paper in Science 16 called for cognitive rehabilitation to be part of the health system response to Long COVID, but rehabilitation was not included in the category of research needs - i.e., the paper implied that investigators already know how to treat patients with PCCS, and that investigators just need to increase access to therapy. However, it is unclear if standard cognitive rehabilitation methods used for other patient groups are effective for people with PCCS. One source of guidance for PCCS rehabilitation methods is the literature on cognitive rehabilitation for adults with traumatic brain injury (TBI), especially patients with mild TBI (aka concussion). Adults with mild TBI (mTBI) have symptoms that are commonly reported by adults with PCCS, such as word-finding problems, slow thinking, "brain fog", trouble following instructions, forgetting medications, difficulty in conversations, complaints about mental fatigue, and difficulty making decisions. There also is anecdotal evidence from clinicians who have overseen treatment of more than 3400 adults with Long COVID - that PCCS characteristics are very similar to patients with mild TBI. COVID and TBI share pathophysiological features such as inflammation, hypoxia, microvascular lesions and disruption of the blood-brain barrier, cortical thinning, and diffuse white-matter damage, particularly in anterior cortical regions. Best practices in cognitive rehabilitation also should be similar in both groups: treatments must be tailored to the patients needs, focused on solving everyday thinking challenges rather than 'fixing' deficits, and given in a relatively high dose.

In summary, PCCS is prevalent, debilitating, and persistent, and there is a lack of evidence-based methods to treat adults with these problems. TBI and COVID share pathophysiological features, survivors report similar cognitive symptoms, and best practices apply to both populations, thus the investigators predict that cognitive rehabilitation methods developed for adults with mTBI will also be effective for adults with PCCS.

Study design will follow recommendations in the CONSORT extension for randomized pilot and feasibility trials, so that data from the Vanguard study can be used in the main trial analysis. Results of the main study will significantly advance the investigators understanding of health consequences of COVID-19, delivery of health care, and health outcomes for adults with Long COVID. It is interdisciplinary research by a Canadian-led research team representing speech-language pathology, occupational therapy, physiotherapy, healthcare administration, and stakeholders with lived experience; and includes US collaborators representing the largest national company providing a cognitive rehabilitation program developed specifically for adults with Long COVID. The investigators collaboration with US partners is a step toward globalization of the rehabilitation methods.

The investigators propose to complete a Vanguard two-arm RCT of STAR-C3 with 100 adults randomized to either Therapy (n=50) or Education (n=50) groups. The study aims to demonstrate the acceptability, appropriateness, and feasibility of STAR-C3 as judged by clinicians and participants with PCCS. Therapy will be delivered by an Occupational Therapist (OT) or Speech-Language Pathologist (SLP).

ELIGIBILITY:
Inclusion Criteria:

* Is a community-dwelling adults
* Is age 18 years or older
* Self-identifies as a fluent English speaker
* Have a history of COVID symptoms as listed on the Government of Canada COVID information website, a positive antigen or polymerase chain reaction (PCR) test, or both
* Have cognitive symptoms that have persisted a minimum of 12 weeks after contracting COVID
* Have cognitive symptoms attributable to COVID and not to other intervening diagnoses associated with cognitive dysfunction (e.g., psychosis, concussion), or medications with negative effects on cognitive function
* Have no previous history of a diagnosis of a neurological disorder affecting thinking (e.g., dementia)
* Are able to participate in 3 one-hour sessions per week for 4-6 weeks
* Are not in active behavioural treatment for a substance-use or mental-health disorder, or in cognitive rehabilitation provided by a registered health professional (e.g., speech-language pathologist or occupational therapist)
* Can access an electronic device with internet access and capability for Zoom videoconferencing

Exclusion Criteria:

* A score of less than 20 on the Montreal Cognitive Assessment (MoCA), which indicates a risk for dementia.
* Cannot identify at least 3 problems on the Common Cognitive Complaints after Concussion Questionnaire (C4), as there would be insufficient areas for intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 9 months
  The primary outcome is the rate of recruitment, average 5 per month. The primary outcome is the rate of recruitment and retention rate reported as the total number of participants recruited and retained.

SECONDARY OUTCOMES:
Acceptability of the Intervention | Measures administered during intake (baseline), immediately after one of sessions 6-10 depending on targets achieved, and 1 month post-treatment.
  The acceptability will be assessed by clinicians and participants. At least three quarters of participants and clinicians will provide a rating of 4 on the Acceptability of Intervention Measure (AIM).
Acceptability of the Appropriateness | Measures administered during intake (baseline), immediately after one of sessions 6-10 depending on targets achieved, and 1 month post-treatment.
  The acceptability will be assessed by clinicians and participants. At least three quarters of participants and clinicians will provide a rating of 4 on the Intervention Appropriateness Measure (IAM).
Acceptability of the Feasibility | Measures administered during intake (baseline), immediately after one of sessions 6-10 depending on targets achieved, and 1 month post-treatment
  The acceptability will be assessed by clinicians and participants. At least three quarters of participants and clinicians will provide a rating of 4 on the Feasibility of Intervention Measure (FIM).

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Bosch, PhD, Principal Investigator — McMaster University School of Rehabilitation Science; Lyn Turkstra, PhD, Principal Investigator — McMaster University School of Rehabilitation Science
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Background] Hampshire A, Trender W, Chamberlain SR, Jolly AE, Grant JE, Patrick F, Mazibuko N, Williams SC, Barnby JM, Hellyer P, Mehta MA. Cognitive deficits in people who have recovered from COVID-19. EClinicalMedicine. 2021 Sep;39:101044. doi: 10.1016/j.eclinm.2021.101044. Epub 2021 Jul 23. PMID 34316551
- [Background] Liu YH, Chen Y, Wang QH, Wang LR, Jiang L, Yang Y, Chen X, Li Y, Cen Y, Xu C, Zhu J, Li W, Wang YR, Zhang LL, Liu J, Xu ZQ, Wang YJ. One-Year Trajectory of Cognitive Changes in Older Survivors of COVID-19 in Wuhan, China: A Longitudinal Cohort Study. JAMA Neurol. 2022 May 1;79(5):509-517. doi: 10.1001/jamaneurol.2022.0461. PMID 35258587
- [Background] Carazo S, Skowronski DM, Laforce R Jr, Talbot D, Falcone EL, Laliberte D, Denis G, Deshaies P, Hegg-Deloye S, De Serres G. Physical, Psychological, and Cognitive Profile of Post-COVID Conditions in Healthcare Workers, Quebec, Canada. Open Forum Infect Dis. 2022 Aug 1;9(8):ofac386. doi: 10.1093/ofid/ofac386. eCollection 2022 Aug. PMID 35983264
- [Background] Ziauddeen N, Gurdasani D, O'Hara ME, Hastie C, Roderick P, Yao G, Alwan NA. Characteristics and impact of Long Covid: Findings from an online survey. PLoS One. 2022 Mar 8;17(3):e0264331. doi: 10.1371/journal.pone.0264331. eCollection 2022. PMID 35259179
- [Background] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Background] Wang C, Han J. Will the COVID-19 pandemic end with the Delta and Omicron variants? Environ Chem Lett. 2022;20(4):2215-2225. doi: 10.1007/s10311-021-01369-7. Epub 2022 Jan 15. No abstract available. PMID 35069059
- [Background] Katzourakis A. COVID-19: endemic doesn't mean harmless. Nature. 2022 Jan;601(7894):485. doi: 10.1038/d41586-022-00155-x. No abstract available. PMID 35075305
- [Background] Gosse PJ, Kassardjian CD, Masellis M, Mitchell SB. Virtual care for patients with Alzheimer disease and related dementias during the COVID-19 era and beyond. CMAJ. 2021 Mar 15;193(11):E371-E377. doi: 10.1503/cmaj.201938. No abstract available. PMID 33722828
- [Background] Chuang HJ, Hsiao MY, Wang TG, Liang HW. A multi-disciplinary rehabilitation approach for people surviving severe COVID-19-a case series and literature review. J Formos Med Assoc. 2022 Dec;121(12):2408-2415. doi: 10.1016/j.jfma.2022.02.002. Epub 2022 Feb 14. PMID 35216882
- [Background] Wise J. Long covid: WHO calls on countries to offer patients more rehabilitation. BMJ. 2021 Feb 10;372:n405. doi: 10.1136/bmj.n405. No abstract available. PMID 33568362
- [Background] Carson G; Long Covid Forum Group. Research priorities for Long Covid: refined through an international multi-stakeholder forum. BMC Med. 2021 Mar 31;19(1):84. doi: 10.1186/s12916-021-01947-0. No abstract available. PMID 33785027
- [Background] Ramage AE. Potential for Cognitive Communication Impairment in COVID-19 Survivors: A Call to Action for Speech-Language Pathologists. Am J Speech Lang Pathol. 2020 Nov 12;29(4):1821-1832. doi: 10.1044/2020_AJSLP-20-00147. Epub 2020 Sep 18. PMID 32946270
- [Background] Alwan NA. The road to addressing Long Covid. Science. 2021 Jul 30;373(6554):491-493. doi: 10.1126/science.abg7113. No abstract available. PMID 34326224
- [Background] Soble JR, Silva MA, Vanderploeg RD, Curtiss G, Belanger HG, Donnell AJ, Scott SG. Normative Data for the Neurobehavioral Symptom Inventory (NSI) and post-concussion symptom profiles among TBI, PTSD, and nonclinical samples. Clin Neuropsychol. 2014;28(4):614-32. doi: 10.1080/13854046.2014.894576. Epub 2014 Mar 14. PMID 24625213
- [Background] Ahman S, Saveman BI, Styrke J, Bjornstig U, Stalnacke BM. Long-term follow-up of patients with mild traumatic brain injury: a mixed-method study. J Rehabil Med. 2013 Sep;45(8):758-64. doi: 10.2340/16501977-1182. PMID 24002311
- [Background] Cancelliere C, Hincapie CA, Keightley M, Godbolt AK, Cote P, Kristman VL, Stalnacke BM, Carroll LJ, Hung R, Borg J, Nygren-de Boussard C, Coronado VG, Donovan J, Cassidy JD. Systematic review of prognosis and return to play after sport concussion: results of the International Collaboration on Mild Traumatic Brain Injury Prognosis. Arch Phys Med Rehabil. 2014 Mar;95(3 Suppl):S210-29. doi: 10.1016/j.apmr.2013.06.035. PMID 24581907
- [Background] Qin Y, Wu J, Chen T, Li J, Zhang G, Wu D, Zhou Y, Zheng N, Cai A, Ning Q, Manyande A, Xu F, Wang J, Zhu W. Long-term microstructure and cerebral blood flow changes in patients recovered from COVID-19 without neurological manifestations. J Clin Invest. 2021 Apr 15;131(8):e147329. doi: 10.1172/JCI147329. PMID 33630760
- [Background] Egbert AR, Cankurtaran S, Karpiak S. Brain abnormalities in COVID-19 acute/subacute phase: A rapid systematic review. Brain Behav Immun. 2020 Oct;89:543-554. doi: 10.1016/j.bbi.2020.07.014. Epub 2020 Jul 17. PMID 32682993
- [Background] Togher L, Wiseman-Hakes C, Douglas J, Stergiou-Kita M, Ponsford J, Teasell R, Bayley M, Turkstra LS; INCOG Expert Panel. INCOG recommendations for management of cognition following traumatic brain injury, part IV: cognitive communication. J Head Trauma Rehabil. 2014 Jul-Aug;29(4):353-68. doi: 10.1097/HTR.0000000000000071. PMID 24984097
- [Background] Tate R, Kennedy M, Ponsford J, Douglas J, Velikonja D, Bayley M, Stergiou-Kita M. INCOG recommendations for management of cognition following traumatic brain injury, part III: executive function and self-awareness. J Head Trauma Rehabil. 2014 Jul-Aug;29(4):338-52. doi: 10.1097/HTR.0000000000000068. PMID 24984096
- [Background] Velikonja D, Tate R, Ponsford J, McIntyre A, Janzen S, Bayley M; INCOG Expert Panel. INCOG recommendations for management of cognition following traumatic brain injury, part V: memory. J Head Trauma Rehabil. 2014 Jul-Aug;29(4):369-86. doi: 10.1097/HTR.0000000000000069. PMID 24984098
- [Background] Ponsford J, Bayley M, Wiseman-Hakes C, Togher L, Velikonja D, McIntyre A, Janzen S, Tate R; INCOG Expert Panel. INCOG recommendations for management of cognition following traumatic brain injury, part II: attention and information processing speed. J Head Trauma Rehabil. 2014 Jul-Aug;29(4):321-37. doi: 10.1097/HTR.0000000000000072. PMID 24984095
- [Background] Tavel JA, Fosdick L; ESPRIT Vanguard Group. ESPRIT Executive Committee. Closeout of four phase II Vanguard trials and patient rollover into a large international phase III HIV clinical endpoint trial. Control Clin Trials. 2001 Feb;22(1):42-8. doi: 10.1016/s0197-2456(00)00114-8. PMID 11165422
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Solianik R, Mickeviciene D, Zlibinaite L, Cekanauskaite A. Tai chi improves psychoemotional state, cognition, and motor learning in older adults during the COVID-19 pandemic. Exp Gerontol. 2021 Jul 15;150:111363. doi: 10.1016/j.exger.2021.111363. Epub 2021 Apr 19. PMID 33887380
- [Background] Daynes E, Gerlis C, Chaplin E, Gardiner N, Singh SJ. Early experiences of rehabilitation for individuals post-COVID to improve fatigue, breathlessness exercise capacity and cognition - A cohort study. Chron Respir Dis. 2021 Jan-Dec;18:14799731211015691. doi: 10.1177/14799731211015691. PMID 33957805
- [Background] Ladds E, Rushforth A, Wieringa S, Taylor S, Rayner C, Husain L, Greenhalgh T. Persistent symptoms after Covid-19: qualitative study of 114 "long Covid" patients and draft quality principles for services. BMC Health Serv Res. 2020 Dec 20;20(1):1144. doi: 10.1186/s12913-020-06001-y. PMID 33342437
- [Background] Hart T, Dijkers MP, Whyte J, Turkstra LS, Zanca JM, Packel A, Van Stan JH, Ferraro M, Chen C. A Theory-Driven System for the Specification of Rehabilitation Treatments. Arch Phys Med Rehabil. 2019 Jan;100(1):172-180. doi: 10.1016/j.apmr.2018.09.109. Epub 2018 Sep 27. PMID 30267669
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Malec JF, Smigielski JS, DePompolo RW. Goal attainment scaling and outcome measurement in postacute brain injury rehabilitation. Arch Phys Med Rehabil. 1991 Feb;72(2):138-43. PMID 1991015
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Kendrick D, Silverberg ND, Barlow S, Miller WC, Moffat J. Acquired brain injury self-management programme: a pilot study. Brain Inj. 2012;26(10):1243-9. doi: 10.3109/02699052.2012.672787. Epub 2012 Jun 1. PMID 22658076
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Nordhues HC, Bhagra A, Stroud NN, Vencill JA, Kuhle CL. COVID-19 Gender Disparities and Mitigation Recommendations: A Narrative Review. Mayo Clin Proc. 2021 Jul;96(7):1907-1920. doi: 10.1016/j.mayocp.2021.04.009. Epub 2021 Apr 20. PMID 34218863
- [Background] Liu N, Zhang F, Wei C, Jia Y, Shang Z, Sun L, Wu L, Sun Z, Zhou Y, Wang Y, Liu W. Prevalence and predictors of PTSS during COVID-19 outbreak in China hardest-hit areas: Gender differences matter. Psychiatry Res. 2020 May;287:112921. doi: 10.1016/j.psychres.2020.112921. Epub 2020 Mar 16. PMID 32240896
- [Background] Landivar LC, Ruppanner L, Scarborough WJ, Collins C. Early Signs Indicate That COVID-19 Is Exacerbating Gender Inequality in the Labor Force. Socius. 2020 Aug 3;6:2378023120947997. doi: 10.1177/2378023120947997. eCollection 2020. PMID 34192138
- [Background] Bowleg L, Landers S. The Need for COVID-19 LGBTQ-Specific Data. Am J Public Health. 2021 Sep;111(9):1604-1605. doi: 10.2105/AJPH.2021.306463. Epub 2021 Aug 26. No abstract available. PMID 34436923
- [Background] Martin S, Mooruth D, Guerdoux-Ninot E, Mazzocco C, Brouillet D, Taconnat L, Trouillet R. Demographic Characteristics, Motivation and Perception of Change as Determinants of Memory Compensation Self-Reports After Acquired Brain Injury. Front Psychol. 2021 Jul 14;12:607035. doi: 10.3389/fpsyg.2021.607035. eCollection 2021. PMID 34335350
- See also: Viral Neuro Exploration (VINEx), COVID Long Haulers Support Group Canada, Neurological Health Charities Canada. Report on Long COVID Impact Survey. 2021 — https://imgix.cosmicjs.com/d8d3d3b0-c936-11eb-ba89-e7f98c8c358b-FINAL---Report-on-Long-Covid-Impact-Survey---June-8-2021.pdf
- See also: Office for National Statistics. Prevalence of ongoing symptoms following coronavirus (COVID-19) infection in the United Kingdom — https://www.ons.gov.uk/peoplepopulationandcommunity/healthandsocialcare/conditionsanddiseases/bulletins/prevalenceofongoingsymptomsfollowingcoronaviruscovid19infectionintheuk/5august2021
- See also: How does COVID-19 affect the brain? A troubling picture emerges. — https://www.nationalgeographic.com/science/article/how-does-covid-19-affect-the-brain-a-troubling-picture-emerges